CLINICAL TRIAL: NCT01924832
Title: Study to Investigate the Pharmacokinetics, Safety, and Tolerability of BG00012 (Dimethyl Fumarate) When Delivered to Different Regions of the Gastrointestinal Tract in Healthy Subjects
Brief Title: BG00012 Regional Absorption Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 109HV111; EUDRA CT NO: 2013-002048-96
Record Dates: First submitted 2013-08-01; First posted 2013-08-19 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
MeSH Terms: interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BG00012 Part 1 (Experimental): BG00012 120 mg delivered to varying locations of the GI tract
  Interventions: Drug: dimethyl fumarate
- BG00012 Part 2 (Experimental): BG00012 240 mg delivered to varying locations of the GI tract
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — tablet
  Other Names: DMF; Tecfidera; BG00012

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics (PK) profile of monomethyl fumarate (MMF) following delivery of BG00012 (dimethyl fumarate, DMF) 120 mg (Part 1) and BG00012 240 mg (Part 2) to varying regions within the GI tract in healthy volunteers. The secondary objective of this study is to evaluate the safety and tolerability profile following the delivery of BG00012 120 mg (Part 1) and BG00012 240 mg (Part 2) to varying regions within the GI tract in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females.
* Body mass index (BMI) of 18 through 35 kg/m2.
* Subjects of childbearing potential (including males) must practice effective contraception during the study and be willing and able to continue contraception for 90 days after their last dose of study treatment

Key Exclusion Criteria:

* History of or positive test result at Screening for human immunodeficiency virus (HIV), hepatitis C virus (HCV) antibody, or hepatitis B virus (defined as positive for hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb]).
* Serious infection (e.g., pneumonia, septicemia) within the 3 months prior to first dose.
* Vaccinations within 4 weeks prior to first dose.
* History of drug or alcohol abuse (as defined by the Investigator) within the previous 2 years, or regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint of beer, 25 mL of 40% spirit or a 125 mL glass of wine).
* History of clinically significant gastrointestinal (GI) disease as determined by the Investigator (including Crohn's Disease, Ulcerative Colitis, confirmed diagnosis of active Irritable Bowel Syndrome).
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The maximum observed concentration: Cmax | Up to week 9
The time to reach maximum observed concentration: Tmax | Up to week 9
The area under the plasma concentration versus time curve from time zero to 24 hours | Up to week 9
The area under the plasma concentration versus time curve from time zero to time t (the last sampling time with quantifiable monomethyl fumarate [MMF]) | Up to week 9
The area under the plasma concentration versus time curve from time zero to infinity | Up to week 9
The apparent elimination half-life | Up to week 9
The time prior to the first quantifiable monomethyl fumarate (MMF) plasma concentration | Up to week 9
Area under the plasma concentration versus time curve (AUC) ratio of test regimens compared with reference for Part 1 | Up to week 9
Area under the plasma concentration versus time curve (AUC) ratio of test regimens compared with reference for Part 2 | Up to week 9

SECONDARY OUTCOMES:
The number of participants that experience Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to week 9

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Nottingham, United Kingdom